CLINICAL TRIAL: NCT02155062
Title: Urinary Alkylresorcinol Metabolites as a Biomarker of Whole Grain Wheat and Rye Intake
Brief Title: Biomarkers of Whole Grain Wheat and Rye Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Julia Darzi, Lecturer Nutrition and Dietetics, King's College London
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BDM/13/14-78
Record Dates: First submitted 2014-05-29; First posted 2014-06-04 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Volunteers
Keywords: Nutritional biomarker; Dietary assessment; Whole grain; Wheat; Rye; Alkylresorcinol; Urine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Whole grain rye (Experimental): 3-4 portions per day of WG rye containing foods (approximately 20 WG per portion)
  Interventions: Other: Whole grain rye; Other: Refined cereal
- Whole grain wheat (Experimental): 3-4 portions per day of WG wheat containing foods (approximately 20 WG per portion)
  Interventions: Other: Whole grain wheat; Other: Refined cereal
- Refined cereal (Placebo Comparator): No intake of WG wheat or WG rye cereals, only refined cereals or non-AR containing WG cereals (e.g. WG rice or oats)
  Interventions: Other: Refined cereal

INTERVENTIONS:
Other: Whole grain rye
  Arms: Whole grain rye
Other: Whole grain wheat
  Arms: Whole grain wheat
Other: Refined cereal

SUMMARY:
Alkylresorcinols (AR) are a group of lipids found in the bran fraction of wheat and rye grains. AR are absorbed into the bloodstream and their metabolites are excreted in urine in measurable amounts following ingestion of wholegrain (WG) wheat or rye cereal. As AR are absent in refined cereals, plasma AR and urinary AR metabolites are proposed as suitable biomarkers of dietary intake of WG wheat and rye cereal, with a number of studies supporting this proposal. Different AR species are present in characteristic quantities in WG wheat in comparison to WG rye cereals, which can allow identification of the main source of WG (wheat or rye) in individuals by analysing the AR concentrations in blood. However the patterns of urinary AR metabolite excretion following wheat or rye intake have not yet been investigated to determine if there are differences according to WG source.

The present study aims to:

(i) investigate the differences in AR metabolite excretion pattern in spot and 24 hour urine samples after following a predominantly WG rye-based diet in comparison to a predominantly WG wheat-based diet and in comparison to control (refined cereal diet) (ii) compare the validity and reproducibility of AR metabolites in spot urine samples in comparison to 24 hour urine samples.

ELIGIBILITY:
Inclusion Criteria:

* Body mass intake 18.5-30.0 kg/m2
* Weight stable for 2 months
* Generally healthy

Exclusion Criteria:

* Previous or current chronic disease including heart disease, diabetes, gastrointestinal, liver, renal or endocrine disorders
* Drug or alcohol misuse in the last year
* Current pregnancy or lactation
* Weight change of >3 kg in the last two months
* Current regular user of certain prescription medications (except contraceptives)
* Unwilling to consume or to stop consuming WG wheat, WG rye or refined cereals
* Unwilling to discontinue multivitamins/dietary supplements during study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
24-h urinary DHBA:DHPPA ratio | Endpoint (Day 3)
  DHBA: 3,5-dihydroxybenzoic acid DHPPA: 3-(3,5-dihydroxyphenyl)-propanoic acid
  DHBA & DHPPA are the main AR metabolites excreted in urine

SECONDARY OUTCOMES:
DHBA:DHPPA ratio in morning spot urine | Endpoint (Day 3)
Total 24-h urinary AR metabolite (DHBA + DHPPA) excretion | Endpoint (Day 3)
Total 24-h urinary DHBA excretion | Endpoint (Day 3)
Total 24-h urinary DHPPA excretion | Endpoint (Day 3)
24-h urinary total AR (DHBA+DHPPA):creatinine ratio | Endpoint (Day 3)
24-h urinary DHBA:creatinine ratio | Endpoint (Day 3)
24-h urinary DHPPA:creatinine ratio | Endpoint (Day 3)
Total AR (DHBA+DHPPA):creatinine ratio in morning spot urine sample | Endpoint (Day 3)
DHBA:creatinine ratio in morning spot urine sample | Endpoint (Day 3)
DHPPA:creatinine ratio in morning spot urine sample | Endpoint (Day 3)

OTHER OUTCOMES:
Estimated daily intake of WG wheat and rye cereals | Assessed throughout each intervention period (Days 1-3)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Darzi, PhD, Principal Investigator — King's College London
Locations (1):
- Diabetes and Nutritional Sciences Division, King's College London, London, United Kingdom